CLINICAL TRIAL: NCT03208829
Title: Effects of an Exercise Program Based on Muscle Strengthening in the Rehabilitation of Individuals Undergoing Total Hip Arthroplasty: a Randomized Clinical Trial.
Brief Title: Exercises in the Post-operative Rehabilitation of THA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Bruna de Moraes Lopes, Principal Investigator (PhD student), Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: THA Rehabilitation
Record Dates: First submitted 2017-07-01; First posted 2017-07-06 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Patients with total hip arthroplasty, will be assigned to two different treatment groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: The random allocation step will be conducted through Randomizers - www.random.org by a research assistant. The assistant responsible for randomization will not be involved in any other phase of the study and the secrecy of the allocation will be maintained through opaque envelopes. A second independent assistant will administer the agenda and all communication between the participants and the researchers involved
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Rehabilitation Exercises Group 1 will be submitted to an exercise protocol based on muscle strength training, with duration of 6 weeks and frequency of two weekly sessions, lasting 45 minutes.
  Interventions: Other: Rehabilitation exercises
- Group 2 (Active Comparator): Postoperative guidance Group 2 will receive an orientation booklet and weekly links from researchers to address possible questions.
  Interventions: Other: Postoperative guidance

INTERVENTIONS:
Other: Rehabilitation exercises — Patients in group 1 will participate in a physical exercise protocol supervised by a physiotherapist. The sessions will focus on the rehabilitation of muscle strength and the exercises will be performed with increased external load.
  Arms: Group 1
Other: Postoperative guidance — Group 2 will receive only guidelines regarding postoperative care.
  Arms: Group 2

SUMMARY:
Subjects submitted to unilateral THA will be randomized into two rehabilitation groups. One group will receive a booklet with guidelines for postoperative care, while the other group will participate in face-to-face sessions with exercises with emphasis on muscle strengthening.

DETAILED DESCRIPTION:
Individuals with osteoarthritis (OA) of the hip submitted to total hip arthroplasty (THA) may present alterations in their functional capacity, and associated, among other aspects, the reduction in muscle strength. Our overall objective is to compare the effects of an exercise program based on training of muscular strength to orientations and functional home exercises in patients submitted to THA, as well as to compare the outcomes of both groups with those of healthy individuals. Individuals with THA will be randomly assigned to two groups. One group will receive face-to-face treatment (G1) and the other will receive postoperative guidance (G2). A blinded appraiser regarding the allocation will apply the evaluation tools at the moments: preintervention, after completing 7 days and after 10 weeks of the end of the treatment. The research will present as clinical outcomes: the muscular strength, through the values of torque peaks obtained in dynamometry; the functional capacity through the results of the Timed Up and Go test and the Harris Hip Score questionnaire; the range of joint motion measured with and flexometer; the pain through the results of the numerical scale of pain; and kinesiophobia, through the scores obtained in the Tampa Scale.

ELIGIBILITY:
Inclusion Criteria:

* Referred by orthopedic doctors of the city of Porto Alegre, Rio Grande do Sul, Brazil;
* Between 30-60 days of unilateral total hip arthroplasty (cemented and hybrid prostheses) postoperative phase;
* Read and consent to the Free and Informed Consent Form and understood the guidelines necessary to carry out the evaluations proposed in this research.

Exclusion Criteria:

* Performing a surgical procedure, in the last six months, in other articular joints in the lower limbs;
* previous surgical procedures in the coxofemoral joint;
* surgical procedures and osteoarticular diseases in the lumbar spine;
* osteoarticular diseases in lower limb joints;
* muscle injuries in lower limbs;
* presence of signs or symptoms of osteoarthritis in the contralateral hip;
* postoperative complications such as prosthesis dislocation, deep venous thrombosis, periarticular fractures and neural lesions;
* intra-articular injection of corticosteroids in the lower limbs during the last six months;
* cardiovascular diseases with presence of disability, such as severe dyspnea and uncontrolled arterial hypertension;
* presence of neurological diseases.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2018-05-04 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
6 Weeks Post-Intervention Muscle Strength | Will be measured post intervention 6 weeks after intervention).
  Muscle strength will be measured by a portable dynamometer and represented as muscle torque (N.m).

SECONDARY OUTCOMES:
Functional Capacity (TUG) | Will be measured pre-intervention (30 days after the surgery), and two moments post intervention (1 week after intervention and 6 weeks after intervention).
  Functional capacity will be evaluated through the timed up and go test.
Functional Capacity (HHS) | Will be measured pre-intervention (30 days after the surgery), and two moments post intervention (1 week after intervention and 6 weeks after intervention).
  Functional capacity will be evaluated through the harris hip score questionnaire.
Hip Range of Motion | Will be measured pre-intervention (30 days after the surgery), and two moments post intervention (1 week after intervention and 6 weeks after intervention).
  Hip range of motion will be measured with a flexometer and presented in degrees of movement.
Pain in the operated hip (last seven days) | Will be measured pre-intervention (30 days after the surgery), and two moments post intervention (1 week after intervention and 6 weeks after intervention).
  The patient will be asked about pain felt in the operated hip within the last 7 days. Pain will be assessed with the numeric pain scale and will be represented by the number selected by the patient.
1 Week Post-Intervention Muscle Strength | Will be measured post intervention (1 week after intervention).
  Muscle strength will be measured by a portable dynamometer and represented as muscle torque (N.m).
Pre-Intervention Muscle Strength | Will be measured pre-intervention (30 days after the surgery).
  Muscle strength will be measured by a portable dynamometer and represented as muscle torque (N.m)

OTHER OUTCOMES:
Body Mass Index | Will be measured pre-intervention (30 days after the surgery), and two moments post intervention (1 week after intervention and 6 weeks after intervention).
  Body mass index will be acquired by measuring weight and height, and presented in form of the equation mass/height².
Length of Lower Limbs | Will be measured pre-intervention (30 days after the surgery), and two moments post intervention (1 week after intervention and 6 weeks after intervention).
  Length of lower limbs will be performed through a tape measure and presented in centimeters.
Kinesiophobia | Will be measured pre-intervention (30 days after the surgery), and two moments post intervention (1 week after intervention and 6 weeks after intervention).
  For the evaluation of the kinesiophobia will be used the Tampa Scale.
Femoral Offset | Will be measured pre-intervention (30 days after the surgery), and two moments post intervention (1 week after intervention and 6 weeks after intervention).
  Evaluation of femoral vertical and horizontal offset, using radiography exams.

CONTACTS AND LOCATIONS:
Overall Officials: Bruna M Lopes, PhD Student, Principal Investigator — Federal Health Science University of Porto Alegre
Locations (1):
- Federal Health Science University of Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No